CLINICAL TRIAL: NCT00754546
Title: Effects of Arformoterol on Exercise Endurance Time and Breathlessness in COPD: Cycle Ergometer vs. Treadmill
Brief Title: Effect of Bronchodilation on Cycle vs Treadmill Exercise Endurance Time in COPD
Acronym: ARFEET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21261
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Results first posted 2013-05-29 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: exercise;; treadmill;; cycle ergometer;; breathlessness;; leg discomfort
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity; Dyspnea | interventions — Formoterol Fumarate; Plyometric Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arformoterol tartrate (Active Comparator): Bronchodilator therapy with arformoterol solution 15 mcg
  Interventions: Drug: Arformoterol tartrate; Other: Treadmill Exercise; Other: Cycle Exercise
- Normal saline (Placebo Comparator): Placebo using normal saline
  Interventions: Drug: Placebo: Normal Saline; Other: Treadmill Exercise; Other: Cycle Exercise

INTERVENTIONS:
Drug: Arformoterol tartrate — 15 mcg in two ml solution administered via nebulizer
  Other Names: Brovana
  Arms: Arformoterol tartrate
Drug: Placebo: Normal Saline — Normal saline was nebulized.
  Arms: Normal saline
Other: Treadmill Exercise
Other: Cycle Exercise

SUMMARY:
Previous studies suggest that treadmill exercise may be a more relevant exercise stimulus than the cycle ergometer to demonstrate benefits with bronchodilator therapy in patients with COPD. The hypothesis of the study is that patients with COPD will exhibit greater improvements in exercise endurance and breathlessness with arformoterol compared with normal saline during treadmill walking than with cycle exercise.

DETAILED DESCRIPTION:
The study is a randomized trial with crossover of consecutively recruited patients with symptomatic COPD. Each patient will participate in seven visits over a 3-4 week period. At the first visit patients will provide informed consent and then be familiarized with equipment and testing protocols. At visits 2 and 3 patients will inhale 2 puffs of albuterol HFA MDI, and then perform symptom limited incremental exercise on the treadmill or cycle ergometer (randomized order); after a one hour rest, the patient will perform constant work exercise at 80-85% of peak VO2 on the same exercise mode.

At visits 4 - 7, patients will perform PFTs at baseline and at 30 and 120 minutes after inhaling arformoterol or normal saline (randomized order) and then constant work exercise on the treadmill or cycle ergometer (randomized order). Metabolic measurements will be made throughout exercise, and patients will provide continuous ratings of breathlessness and leg discomfort using a system consisting of a computer, monitor, and a mouse.

ELIGIBILITY:
Inclusion Criteria:

* male or female patient 50 years of age or older; diagnosis of COPD; current or ex-smoker with at least 10 pack-years of smoking; a patient-reported score for breathlessness during activities of daily living of < 9 on the self-administered computerized baseline dyspnea index; a post-bronchodilator FEV1 < 80% predicted; a post-bronchodilator FEV1/FVC ratio < 70%; and clinically stable condition.

Exclusion Criteria:

* any concomitant disease that interferes with study procedures or evaluation; inability to exercise on the treadmill or cycle ergometer; inability to withhold short-acting bronchodilators for 4 hours or long-acting bronchodilators for 12 hrs (salmeterol or formoterol) and for 24 hours (tiotropium) prior to testing

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doanld A Mahler, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Result] Zhang X, Waterman LA, Ward J, Baird JC, Mahler DA. Advantages of endurance treadmill walking compared with cycling to assess bronchodilator therapy. Chest. 2010 Jun;137(6):1354-61. doi: 10.1378/chest.09-2470. Epub 2009 Dec 29. PMID 20040610

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from a specialty clinic in Lebanon, NH, between August 1, 2008 to May 1, 2009.
Pre-assignment Details: 27 particpants recruited; 27 particpants screened; 5 excluded because they did not meet inclusion criteria; 2 patients withdrew consent after visit 1.
Groups:
- All Participants: All 20 participants were randomized to receive all 4 of the interventions in a randomzied sequence. The 4 interventions follow:
  Treadmill exercise-Arformoterol Treadmill exercise-Normal Saline Cycle exercise-Arformoterol Cycle exercise-Normal Saline
Period: Overall Study
Arm/Group | All Participants
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 64 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Exercise Endurance Time
Description: Participants were asked to exercise until symptom limitation
Time Frame: After one dose
Population: Number of participants determined by previous studies. Analysis was intention to treat
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Treadmill Exercise With the Active Comparator | Cycle Exercise With the Active Comparator | Treadmill Exercise With the Placebo Comparator | Cycle Exercise With the Placebo Comparator
Number analyzed (Participants) | 20 | 20 | 20 | 20
seconds | 490 (258) | 333 (158) | 472 (258) | 362 (104)
Statistical Analysis 1: Comparison: Treadmill Exercise With the Active Comparator vs Cycle Exercise With the Active Comparator vs Treadmill Exercise With the Placebo Comparator vs Cycle Exercise With the Placebo Comparator; ANOVA was used to examine the interaction between mode of exercise and treatment effect. Twenty patients were considered adequate to provide a power of 85% with an alpha of 0.05; Test type: Superiority or Other; p < 0.05, ANOVA
Statistical Analysis 2: Comparison: Treadmill Exercise With the Active Comparator vs Cycle Exercise With the Active Comparator vs Treadmill Exercise With the Placebo Comparator vs Cycle Exercise With the Placebo Comparator; Comparing arformoterol with placebo with treadmill exercise; Test type: Superiority or Other; p = 0.024, t-test, 2 sided
Statistical Analysis 3: Comparison: Treadmill Exercise With the Active Comparator vs Cycle Exercise With the Active Comparator vs Treadmill Exercise With the Placebo Comparator vs Cycle Exercise With the Placebo Comparator; Arformoterol versus normal saline with cycle exercise; Test type: Superiority or Other; p = 0.038, t-test, 2 sided

2. Secondary Outcome: Linear Regression Between Breathlessness Ratings (on 0 - 10 Borg Scale) and Time Throughout Exercise
Description: linear regression slope of breathlessness - time for arformoterol and for normal saline will be compared between treadmill and cycle exercise
  The higher the number the worse the shortness of breath
Time Frame: After one dose
Measure: Least Squares Mean (Standard Deviation); unit: breathlessness units/min
Arm/Group | Treadmill Exercise With the Active Comparator | Cycle Exercise With the Active Comparator | Treadmill Exercise With the Placebo Comparator | Cycle Exercise With the Placebo Comparator
Number analyzed (Participants) | 20 | 20 | 20 | 20
breathlessness units/min | 1.27 (0.56) | 1.79 (1.05) | 1.42 (0.97) | 1.49 (0.59)

ADVERSE EVENTS:
Arm/Group | Treadmill Exercise With the Active Comparator | Cycle Exercise With the Active Comparator | Treadmill Exercise With the Placebo Comparator | Cycle Exercise With the Placebo Comparator
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
Study completed with no reported adverse effects. One limitation of the study is frequent exercise tests involving 7 visits for each participant

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No